CLINICAL TRIAL: NCT03561779
Title: A Randomized, Double-blind, Active-controlled, Multi-center, Phase 3 Study to Evaluated the Safety and Efficacy of Intraarticular Hyalurinic Acid(YYD302) for Osteoarthritis of the Knee After 12 Weeks of Treatment and Retreatment
Brief Title: Clinical Trial of YYD302 (Phase3) for Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YY_YYD302_003
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The Subjects are injected investigational Product (YYD302 or Synovian Inj.)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYD302 (Experimental): YYD302 (2ml)
  Interventions: Drug: YYD302 2ml
- Synovian Inj. (Active Comparator): Synovian Inj. (3ml)
  Interventions: Drug: Active comparator: Synovian Inj.

INTERVENTIONS:
Drug: YYD302 2ml — YYD302 2ml
  Arms: YYD302
Drug: Active comparator: Synovian Inj. — Active comparator: Synovian Inj.
  Other Names: Synovian Inj.
  Arms: Synovian Inj.

SUMMARY:
This is a randomized, double-blind, active-controlled, multi-center, phase 3 study to evaluate the safety and efficacy of intraarticular hyaluronic acid(YYD302) for osteoarthritis of the knee after 12 weeks of treatment and retreatment

DETAILED DESCRIPTION:
First Injection: A multicenter, active-controlled, randomized, evaluator and subject bllinded, parallel, phase 3 study Re-Injection: A multicenter, active-controlled, randomized, parallel

ELIGIBILITY:
Inclusion Criteria:

[Visit 1, 2 Inclusion Criteria]

1. Males or Females 40 years and older
2. According to the clinical diagnosis standard of the American College of Rheumatology (ACR), someone, diagnosed as a single/both sides of osteoarthritis, who corresponds to over 3 conditions of followings.

1) Over 50 years of age 2) Less than 30 minutes of morning stiffness 3) Crepitus on active motion 4) 4 bony tenderness 5) Bony enlargement 6) Nopalpable warmth of synvium 3. Within 6 months from screening visit, someone who diagnosed with Kellgren & Lawrence Grade I~III by the radioactive examination.

4. By the Weight-bearing pain(100mm-VAS) examination, someone who has a outcome of the single or both sides of the osteoarthritis is over 40mm 5. Patient (No-responder) who has experienced steady pain in spite of dosing NSAIDs or other pain-killers in the past.

6. Patient who can walk by themselves without helper like cane or walker etc. (If the patient who has used helper routinely from previous 6 months, evaluating the patient including the helper is possible. In this case, patient needs to use same helper continuously by end of the clinical trial test.) 7. Patient who agrees to participate in this clinical trial by themselves.

[Visit 6, 7 Inclusion criteria] 1. According to the clinical diagnosis standard of the American College of Rheumatology (ACR), someone, diagnosed as a single/both sides of osteoarthritis, who corresponds to over 3 conditions of followings.

1. Over 50 years of age
2. Less than 30 minutes of morning stiffness
3. Crepitus on active motion
4. 4 bony tenderness
5. Bony enlargement
6. Nopalpable warmth of synvium 2. At Re-screening visit, someone who diagnosed with Kellgren & Lawrence Grade I~III by the radioactive examination.

3. Patient who can walk by themselves without helper like cane or walker etc. (If the patient who has used helper routinely from previous 6 months, evaluating the patient including the helper is possible. In this case, patient needs to use same helper continuously by end of the clinical trial test.) 4. Patient who are confirmed for Responder by efficacy at visit 5.

Exclusion Criteria:

1. Someone who has BMI≥32kg/m² at the screening visit.
2. Patient who has an experience dosing psychoactive drug, narcotic analgesic which can have an effect on pain sense over 3 months habitually.
3. Patient who has been administrated gastrointestinal drug(for example H₂-blockers, misoprostol or proton pump inhibitors) regularly, who can't stop injecting for clinical study period.
4. Patient has attended abnormal values from screening test(2 times excess at upper limit of the normal values at ALT, AST, BUN, Serum Creatinine).
5. Patient who has rheumarthritis or other inflammatory metabolic arthritis.
6. Patients having serious gastrointestinal, liver, renal, heart disease.
7. When the inflammatory disease is occurred on joint area to patient like septic arthritis.
8. Patients having skin ailment at the injecting site of the joint region.
9. Patients having secondary osteoarthritis according to the Ochronosis, Hemochromatosis or systemic disease.
10. Patients who have severe pain like Sudek's atrophy, Paget's disease, Spinal disc herniation.
11. Poly-articular patients who have suffered seriously by osteoarthritis at other parts affect judge of the knee joint pain.
12. Patients who diagnosed clear interval disappearance at the knee joint by X-ray.
13. Patients who were administrated below drugs before baseline visit. 1) Patients who were injected HA at the target knee joint or other parts of knee joint in recent 9 months.

2) Patients who were injected steroids into the intra-articular knee joint in recent 3 months 3) Patients who were administrated steroids systemically by the oral medication (But, except inhalation) 4) Patients who were administerated Osteoarthritis nutrition such as glucosamine/chondroichin sulfate or physical therapy or herbal remedy(acupuncture, yellowish swelling, moxa cautery) for the purpose of pain relief in recent 2 weeks 5) Patients who have administerated steroid/No-steriod NSAIDs or other pain relief drugs (patch or other external medicine) in recents 2 weeks except Acetaminophen or below 300mg/day of Asprin 14. Patients who have joint effusion trouble were judged as a positive by tests like Patella tap test.

15. Patients who have target knee joint gotten surgical operation history including Arthroscopy within past one year (In case of having other side of knee joint or hip joint gotten surgical operation history, excepting the patients if there is possibility which can influence the target knee joint's appraisal.

16. Patients who have an operation history about target knee joint. 17. Patients who do the height weight aerobic exercise or anaerobic exercise. 18. Patients who need to be administrated anticoagulant agent together(But, except 300mg daily dose aspirin) 19. Patients who have hypersensitivity history about Investigational Product.

20. In the midst of women in their childbearing years, patients who disagree to do * contraception by medically permitted method for 12 weeks from administrating investigational product.

* The contraception by medically permitted method: Condom, In case of using injection or insertion, In case of installing a intrauterine contraception device etc.

  21. Pregnant and lactating women 22. Patients who were injected other investigational product over a time within 30 days before participated in this clinical trail.

  23. Besides that, the patients who have difficulty to be participated in this clinical trial continuously by Principle Investigator (PI)'s decision.
* Exclusion criteria for Re-injection is except for 13-1) Re-injection date is followed by visit 7.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of change of the Weight-bearing pain(100mm-VAS) on 12 weeks after first injection in comparison with baseline | Change of the week 12 from baseline
  Weight-bearing pain(100mm-VAS) assessed by the subject

SECONDARY OUTCOMES:
Rate of change of the Weight-bearing pain(100mm-VAS) on 2, 4 weeks after administration in comparison with baseline | Change of the week 2, 4 from baseline
  Weight-bearing pain(100mm-VAS) assessed by the subject
Rate of change of the KOOS scales on the 2, 4, 12 weeks after administration in comparison with baseline | Change of the week 2, 4, 12 from baseline
  KOOS scales assessed by the subject
Rate of change of the rest pain(100mm-VAS) on the 2, 4, 12 weeks after administration in comparison with baseline | Change of the week 2, 4, 12 from baseline
  Rest pain(100mm-VAS) assessed by the subject
Rate of change of the Motion pain (100mm-VAS) on the 2, 4, 12 weeks after administration in comparison with baseline | Change of the week 2, 4, 12 from baseline
  Motion pain(100mm-VAS) assessed by the subject
Patient global assessment (100mm-VAS) on the 2, 4, 12 weeks after administration with baseline | Change of the week 2, 4, 12 from baseline
  Patient global assessment (100mm-VAS) assessed by the subject
Investigator global assessment (100mm-VAS) on the 2, 4, 12 weeks after administration with baseline | Change of the week 2, 4, 12 from baseline
  Patient global assessment (100mm-VAS) assessed by the investigator
Change of the swelling in the knee joint from baseline to 2, 4, 12 weeks after administration | Change of the week 2, 4, 12 from baseline
  Sweeling assessed by the investigator
Change of the tenderness on pressure in the knee joint from baseline to 2, 4, 12 weeks after administration | Change of the week 2, 4, 12 from baseline
  Tenderness on pressure assessed by the investigator
Variation of the Range Of Motion(ROM) in the knee joint on 2, 4, 12 weeks after administration with baseline | Change of the week 2, 4, 12 from baseline
  Range of motion assessed by the investigator
Responder rate of the Weight-bearing pain on 12 weeks in comparison with baseline | Change of the week 12 from baseline
  Responder rate of the Weight-bearing pain assessed by the investigator
Responder rate of the OMERACT-OARSI on 12 weeks in comparison with baseline | Change of the week 12 from baseline
  Responder rate of the OMERACT-OARSI assessed by the investigator
Use of rescue medication count and the total amount on each visit after injection | Change of the each visit(2, 4, 12, 24, 36 weeks) after injection
  Use of rescue medication count and the total amount assessed by subject
The efficacy of secondary outcome 1~11 after 12 weeks(36weeks) compared with the Re-injection(24weeks) in re-injection subjects | Change of the week 12 (36 weeks) after Re-injection(24weeks)
  Each outcome assessed by the investigator or subject
The efficacy of secondary outcome 1~11 after baseline compared with 2, 4, 12, 24, 36 weeks in Re-injection subjects | Change of the week 2, 4, 12, 24, 36 from baseline
  Each outcome assessed by the investigator or subject

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Won Ha, M.D, Principal Investigator — Samsung Medical Center, Department of Internal Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park YG, Ha CW, Yoo JH, Lee WS, Lee HJ, In Y, Bae KC, Shon OJ, Kim YM, Seon JK, Song SJ, Chang CB, Kim JM, Kim CW, Kim DH, Bae JH. Intra-Articular Injection of a Novel DVS Cross-Linked Hyaluronic Acid Manufactured by Biological Fermentation (YYD302) in Patients With Knee Osteoarthritis: A Double-Blind, Randomized, Multicenter, Noninferiority Study. Clin Ther. 2021 Nov;43(11):1843-1860. doi: 10.1016/j.clinthera.2021.09.005. Epub 2021 Nov 1. PMID 34736768